CLINICAL TRIAL: NCT05060731
Title: Intravenous Ferric Carboxymaltose Versus Oral Ferrous Sulfate Replacement in Anaemia Due to Acute Nonvariceal Gastrointestinal Bleeding (FIERCE): Protocol of a Multicentre Randomised Controlled Trial
Brief Title: Iron Supplementation in Upper Non-variceal Gastrointestinal Bleeding
Acronym: FIERCE
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, dr Erőss Bálint, Principal Investigator, Director of the Centre for Translational Medicine at University of Pécs, University of Pecs
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 46395-5/2021/EÜIG
Record Dates: First submitted 2021-09-17; First posted 2021-09-29 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-10

CONDITIONS: GastroIntestinal Bleeding; Anemia
Keywords: non-variceal upper gastrointersinal bleeding; iron supplementation; intravenous iron
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Anemia

STUDY DESIGN:
Intervention Model Description: The investigators plan to recruit 285 patients on each arm.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral iron supplementation (Active Comparator): Patients randomized to receive oral ferrous sulfate, ca. 200-300 mg every day for 3 months.
  Interventions: Drug: Oral iron supplementation
- Intravenous iron supplementation (Active Comparator): Patients randomized to receive one dose of 1000 mg intravenous ferric carboxymaltose.
  Interventions: Drug: Intravenous iron supplementation

INTERVENTIONS:
Drug: Oral iron supplementation — Ca. 200-300 mg of ferrous sulfate will be administered orally every day for 3 months.
  Arms: Oral iron supplementation
Drug: Intravenous iron supplementation — One dose of intravenous 1000 mg ferric carboxymaltose will be administered on the day of randomization.
  Arms: Intravenous iron supplementation

SUMMARY:
Anemia is a frequent complication of gastrointestinal bleeding, affecting 61% of the patients. Currently, anemia caused by gastrointestinal bleeding can be treated with iron supplementation. However, the dose and route of the administration are still a question. The FIERCE clinical trial aims to compare the effect of intravenous iron supplementation and oral iron replacement on mortality, unplanned emergency visits, and hospital readmissions in multimorbid patients with acute nonvariceal gastrointestinal bleeding.

DETAILED DESCRIPTION:
In gastrointestinal bleeding (GIB) iron deficiency anemia (IDA) is a common complication, affecting more than 60% of the patients. There are two pillars of the treatment of acute GIB. First, the bleeding point needs identification and endoscopic treatment. Second, the resulting hypovolemia and anemia require fluid resuscitation, transfusion, and replacement of the lost iron. There are two simple ways to manage IDA after acute GIB. Patients either have intravenous (IV) iron infusions one to six times as part of their hospital treatment or receive three months of oral iron supplementation. There is a gap in current guidelines on which approach clinicians should choose.

Here the investigators plan a multicentric, two-arm, randomized controlled trial, to compare the efficacy of oral and intravenous iron supplementation in multimorbid patients with acute nonvariceal gastrointestinal bleeding. Patients will be randomly allocated in a 1:1 ratio to two groups. Group A will receive one dose of 1000 mg of IV ferric carboxymaltose on the day of randomization, while iron supplementation for group B will be performed with one ferrous sulfate tablet every day (ca. 200-300 mg) for three months. The primary outcome will be the composite outcome of all-cause mortality, unplanned emergency visit, and unplanned hospital readmission within six months after enrollment.

In the first phase, the investigators plan to recruit 15 patients on each arm to assess the proportion of the primary outcome in the two groups. In the second phase, a sample size calculation for the primary outcome will be performed based on the results of the first phase.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 65 years;
2. endoscopically proven acute nonvariceal GIB source;
3. 48 hours after the endoscopic diagnosis and/or treatment;
4. hemodynamically stable;
5. the discharge of the patient is planned;
6. hemoglobin level <10 g/dl on the day of randomisation;
7. 24 hours after the last transfusion and no need for further transfusion;
8. signed informed consent.

Exclusion Criteria:

1. known hypersensitivity to iron products (mild side effects excluded);
2. previous diagnosis of iron overload [e.g., transferrin receptor saturation (TSAT) >50%, ferritin> 160 for women ng/ml, ferritin >270 ng/ml for men) or disorders of iron utilisation;
3. pregnancy or breast feeding;
4. diagnosis of iron malabsorption (at discretion of the attending clinician; e.g., severe inflammatory bowel disease, active celiac disease);
5. chronic end stage diseases (chronic heart failure-New York Heart Association Classification class 4, chronic kidney disease (eGFR <30 mL/min/1.73 m2) with or without dialysis, liver cirrhosis with Child Pugh C score, chronic kidney disease with dialysis, chronic obstructive pulmonary disease stage 4, chronic inflammatory disease, malignancies, AIDS);
6. active malignancies;
7. liver cirrhosis with known varices at high risk of bleeding - endoscopic features of high risk of variceal bleeding or liver stiffness measured by transient elastography >20 kiloPascal and platelet count <150 × 10^9 cells/L;
8. gastrointestinal tract malignancies with high risk of gastrointestinal bleeding;
9. high risk of poor compliance or no fixed abode;
10. myelo- or lymphoproliferative diseases;
11. anemia not attributable to iron deficiency (sideroblastic anaemia, aplastic anaemia, haemolytic anaemia, thalassaemia, B12 vitamin or folic acid deficiency or combination of these with IDA);
12. primary coagulation disorders (e.g. Glanzmann thrombasthenia, Von Willebrand disease, Haemophylia A, Haemophylia B);
13. the patient will be transferred to another institute after discharge (e.g. hospital, senior care center);
14. Eastern Cooperative Oncology Group (ECOG) Performance Status >2.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 570 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Composite outcome | 3 months
  The composite endpoint includes all-cause mortality, unplanned emergency visit (general practitioner or emergency outpatient clinic), and unplanned hospital admission for any reason. The investigators will calculate the proportion of the outcome in each arm.

SECONDARY OUTCOMES:
All-cause mortality | 1, and 3 months
  Death from any cause. The proportion of the outcome will be calculated in each arm and compared between the arms. The investigators will compare subgroups of patients based on the cause of mortality.
Unplanned emergency visits | 1, and 3 months
  Emergency visit from any cause. The proportion of the outcome will be calculated in each arm and compared between the arms. The investigators will compare subgroups of patients based on the cause of unplanned emergency visits.
Unplanned hospital admission | 1, and 3 months
  Hospital admission from any cause. The proportion of the outcome will be calculated in each arm and compared between the arms. The investigators will compare subgroups of patients based on the cause of unplanned admission.
Quality of life using the 36-Item Short-Form Health Survey | 1, and 3 months +/- 7 days
  Changes in quality of life measured with the 36-Item Short-Form Health Survey (SF-36) questionnaire compared to baseline.
Quality of life using the EuroQol five-dimensions - 5 levels questionnare | 1, and 3 months +/- 7 days
  Changes in quality of life measured with the EuroQol five-dimensions - 5 levels (EQ-5D-5L) questionnaire compared to baseline.
Gait speed | 1, and 3 months +/- 7 days
  Changes in gait speed compared to baseline. Gait speed will be evaluated on a 4-meter flat walking path.
Six-Minute Walk Test (6MWT) | 1, and 3 months +/- 7 days
  Changes in Six-Minute Walk Test (6MWT) compared to baseline.
Handgrip strength | 1, and 3 months +/- 7 days
  Changes in handgrip strength compared to baseline.
Normalization of the haemoglobin level | 1, and 3 months +/- 7 days
  The percentage of participants with Hb levels of ≥12 g/dL in women and ≥13 g/d, compared to baseline.
Change in Hb level | 1, and 3 months +/- 7 days
  Absolute change from baseline to follow-up in Hb level.
Change in haematocrit | 1, and 3 months +/- 7 days
  Absolute change from baseline to follow-up in haematocrit.
Change in serum iron level | 1, and 3 months +/- 7 days
  Absolute change from baseline to follow-up in serum iron level.
Change in serum transferrin level | 1, and 3 months +/- 7 days
  Absolute change from baseline to follow-up in serum transferrin level.
Change in transferrin saturation | 1, and 3 months +/- 7 days
  Absolute change from baseline to follow-up in transferrin saturation.
Change in soluble transferrin receptor concentration | 1, and 3 months +/- 7 days
  Absolute change from baseline to follow-up in soluble transferrin receptor (sTfR) concentration.
Change in ferritin level | 1, and 3 months +/- 7 days
  Absolute change from baseline to follow-up in ferritin level.
Change in the number of reticulocytes | 1, and 3 months +/- 7 days
  Absolute change from baseline to follow-up in the number of reticulocytes.
Change in the number of erythrocytes | 1, and 3 months +/- 7 days
  Absolute change from baseline to follow-up in the number of erythrocytes.
Change in the total iron-binding capacity | 1, and 3 months +/- 7 days
  Absolute change from baseline to follow-up in the total iron-binding capacity (TIBC).
Change in erythropoietin level | 1, and 3 months +/- 7 days
  Absolute change from baseline to follow-up in erythropoietin level.
Change in C-reactive protein level | 1, and 3 months +/- 7 days
  Absolute change from baseline to follow-up in the C-reactive protein level.
Change in hepcidin level | 1, and 3 months +/- 7 days
  Absolute change from baseline to follow-up in hepcidin level.
Change in phosphate level | 1, and 3 months +/- 7 days
  Absolute change from baseline to follow-up in phosphate level.
Discontinuation of the treatment due to adverse events | 1, and 3 months +/- 7 days
  The percentage of discontinuation in the two arms.
Cost-effectiveness | 1, and 3 months +/- 7 days
  The incremental cost-effectiveness ratio (ICER): incremental costs divided by incremental effectiveness .

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Translational Medicine, University of Pécs, Pécs, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McNutt MK, Bradford M, Drazen JM, Hanson B, Howard B, Jamieson KH, Kiermer V, Marcus E, Pope BK, Schekman R, Swaminathan S, Stang PJ, Verma IM. Transparency in authors' contributions and responsibilities to promote integrity in scientific publication. Proc Natl Acad Sci U S A. 2018 Mar 13;115(11):2557-2560. doi: 10.1073/pnas.1715374115. Epub 2018 Feb 27. PMID 29487213
- [Background] McLean E, Cogswell M, Egli I, Wojdyla D, de Benoist B. Worldwide prevalence of anaemia, WHO Vitamin and Mineral Nutrition Information System, 1993-2005. Public Health Nutr. 2009 Apr;12(4):444-54. doi: 10.1017/S1368980008002401. Epub 2008 May 23. PMID 18498676
- [Background] Ferrer-Barcelo L, Sanchis Artero L, Sempere Garcia-Arguelles J, Canelles Gamir P, P Gisbert J, Ferrer-Arranz LM, Monzo Gallego A, Plana Campos L, Huguet Malaves JM, Lujan Sanchis M, Ruiz Sanchez L, Barcelo Cerda S, Medina Chulia E. Randomised clinical trial: intravenous vs oral iron for the treatment of anaemia after acute gastrointestinal bleeding. Aliment Pharmacol Ther. 2019 Aug;50(3):258-268. doi: 10.1111/apt.15327. Epub 2019 Jun 14. PMID 31197861
- [Background] Bager P, Dahlerup JF. Randomised clinical trial: oral vs. intravenous iron after upper gastrointestinal haemorrhage--a placebo-controlled study. Aliment Pharmacol Ther. 2014 Jan;39(2):176-87. doi: 10.1111/apt.12556. Epub 2013 Nov 19. PMID 24251969
- [Background] Tolkien Z, Stecher L, Mander AP, Pereira DI, Powell JJ. Ferrous sulfate supplementation causes significant gastrointestinal side-effects in adults: a systematic review and meta-analysis. PLoS One. 2015 Feb 20;10(2):e0117383. doi: 10.1371/journal.pone.0117383. eCollection 2015. PMID 25700159
- [Background] Sultan P, Bampoe S, Shah R, Guo N, Estes J, Stave C, Goodnough LT, Halpern S, Butwick AJ. Oral vs intravenous iron therapy for postpartum anemia: a systematic review and meta-analysis. Am J Obstet Gynecol. 2019 Jul;221(1):19-29.e3. doi: 10.1016/j.ajog.2018.12.016. Epub 2018 Dec 19. PMID 30578747
- [Background] Cotter J, Baldaia C, Ferreira M, Macedo G, Pedroto I. Diagnosis and treatment of iron-deficiency anemia in gastrointestinal bleeding: A systematic review. World J Gastroenterol. 2020 Dec 7;26(45):7242-7257. doi: 10.3748/wjg.v26.i45.7242. PMID 33362380
- [Derived] Teutsch B, Vancsa S, Farkas N, Szakacs Z, Vorhendi N, Boros E, Szabo I, Hagendorn R, Alizadeh H, Hegyi P, Eross B. Intravenous ferric carboxymaltose versus oral ferrous sulfate replacement in elderly patients after acute non-variceal gastrointestinal bleeding (FIERCE): protocol of a multicentre, open-label, randomised controlled trial. BMJ Open. 2023 Mar 14;13(3):e063554. doi: 10.1136/bmjopen-2022-063554. PMID 36918236
- See also: Related Info — https://tm-centre.org/en/research/clinical-trials/